CLINICAL TRIAL: NCT01982006
Title: Impact Médico-Economique de la Chirurgie de la cATaracte au Laser Femtoseconde
Brief Title: Economic Evaluation of Femtosecond Laser Assisted Cataract Surgery
Acronym: FEMCAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUBX 2012/23
Record Dates: First submitted 2013-10-21; First posted 2013-11-13 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Cataract
Keywords: cataract surgery; femtosecond laser cataract surgery; phacoemulsification; Cost-Benefit Analysis; Cost Effectiveness; Hospital Costs
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction; Phacoemulsification

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phaco (Active Comparator): Cataract surgery by phacoemulsification
  Interventions: Procedure: Cataract surgery with Phacoemulsification
- Femto (Experimental): Corneal incision, anterior capsulorhexis and lens fragmentation by femtosecond laser
  Interventions: Device: Femtosecond laser-assisted cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery with Phacoemulsification — Each patients randomized in the phaco arm will undergo a conventional cataract surgery.
  Corneal incisions will be manually performed using the same calibrated blade and at the same location for all procedures of one surgeon.
  Phacoemulsification machine used to perform cataract surgery in each center will be the same for all patients included in the center. The IOL (IntraOcular Lens) used in each center will be the same for all patients treated in the center.
  Arms: Phaco
Device: Femtosecond laser-assisted cataract surgery — Each patients randomized in the femto arm will undergo a femtosecond laser assisted cataract surgery.
  Corneal incisions will be performed by the laser. Number, size and location of the incisions must be the same than in the phaco arm for all patients treated by one surgeon.
  Phacoemulsification machine used to remove the liquefied lens will be the same than in the phaco arm The IOL used in each center will be the same than in the phaco arm
  Arms: Femto

SUMMARY:
Cataract is the leading cause of blindness worldwide and cataract surgery is the most frequent surgery performed in France. A new technology, the femtosecond laser-assisted cataract surgery, has to be compared with phacoemulsification alone, the conventional cataract surgery, to determine the economic impact of femtosecond laser-assisted process for the French healthcare insurance.

DETAILED DESCRIPTION:
An estimated 700,000 cataract procedures are performed every year in France, with this amount of surgeries predicted to climb as the population there, as well as around the world, ages. Currently, phacoemulsification alone is the conventional cataract surgery. The femtosecond laser-assisted cataract surgery has to be compared with the standard process to provide information on how it could benefit the patient population treated every year for cataract surgery. This economic study has received a grant from the French Ministry of Health to evaluate the economic impact of femtosecond laser-assisted process for the French healthcare system. For this goal, this prospective, randomized, parallel, multicenter and simple blind study will determine the incremental cost/effectiveness ratio for femtosecond laser-assisted process versus phacoemulsification surgery. Visual acuity results and intraoperative or postoperative complication rate will be compared between both groups. The learning curve of the femtosecond laser assisted cataract surgery will be also evaluated for each surgeon involved in the study.

Ethic and regulatory autority authorisations were obtained at 19/Dec/2012 and 15/Feb/2013, respectively. Date of first inclusion: 9/Oct/2013. Date of first NCT release: 13/Nov/2013. 30 patients were included between this period. French regulatory process dos not require NCT registration before first inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Cataract with impaired visual acuity (> or equal +0.3 LogMAR) or with cataract-related visual symptoms (Halos, Monocular diplopia, glare)
* French healthcare insurance beneficiary

Exclusion Criteria:

* Pupil size lower than 6mm
* Iris constriction
* Iris synechiae
* Preoperative zonular instability or crystalline lens subluxation
* Obstructive Corneal scars
* Obstructive pterygion
* Axial length <20.5 mm
* Corneal astigmatism >1.5 diopters
* Fuchs corneal dystrophy
* History of Central retinal vein or artery occlusion
* History of uveitis
* History of optic nerve head neuropathy except glaucoma
* Progressive glaucoma
* Nystagmus
* Uncontrolled diabetes mellitus
* General history of dementia or psychotic disorders
* Pregnancy, breast feeding
* General medications: Alpha-blockers, Carbonic anhydrase inhibitors

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 920 (Actual)
Dates: Start 2013-10-09 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Incremental Cost/effectiveness ratio defined as cost per incremental therapeutic success. | 3 months after inclusion
  Therapeutic success will be defined by the association of the following criterion:
  * No severe intraoperative or postoperative complications,
  * Best Corrected Visual Acuity of 0 LogMAR,
  * A refractive error inferior or equal to 0.75 diopter,
  * Corneal surgically-induced astigmatism inferior or equal to 0.5 diopter and a postoperative change of astigmatism axis inferior or equal to 20°.

SECONDARY OUTCOMES:
Quality of life | Before surgery (From day -8 to day -1) and months 1, 3 and 12 after surgery
  Quality of life evaluation using Visual Function 14 questionnaire
Learning curve of the femtosecond laser-assisted cataract surgery | End of research (Month 12)
Overall costs of cataract surgery in both arms from the hospital perspective | End of research (Month 12)
Incremental cost - Utility ratio defined as incremental Cost/QALY (Quality Adjusted Life Year) for healthcare insurance in both arms | 12 months after inclusion
No severe intraoperative or postoperative complications | 3 months after inclusion
Best Corrected Visual Acuity of 0 LogMAR | 3 months after inclusion
Refractive error inferior or equal to 0.75 diopter | 3 months after inclusion
Corneal surgically-induced astigmatism inferior or equal to 0.5 diopter and a postoperative change of astigmatism axis inferior or equal to 20° | 3 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Cédric SCHWEITZER, MD, Principal Investigator — University Hospital Bordeaux, France; BENARD Antoine, MD, Study Chair — University Hospital Bordeaux, France
Locations (5):
- France (5):
  - CHU de Bordeaux, Bordeaux
  - CHU de Brest, Brest
  - Hospices Civils de Lyon, Lyon
  - Hôpital Cochin, Paris
  - CHU de Tours, Tours

REFERENCES:
- [Background] Abraham AG, Condon NG, West Gower E. The new epidemiology of cataract. Ophthalmol Clin North Am. 2006 Dec;19(4):415-25. doi: 10.1016/j.ohc.2006.07.008. PMID 17067897
- [Background] Resnikoff S, Pascolini D, Etya'ale D, Kocur I, Pararajasegaram R, Pokharel GP, Mariotti SP. Global data on visual impairment in the year 2002. Bull World Health Organ. 2004 Nov;82(11):844-51. Epub 2004 Dec 14. PMID 15640920
- [Background] Lamoureux EL, Fenwick E, Pesudovs K, Tan D. The impact of cataract surgery on quality of life. Curr Opin Ophthalmol. 2011 Jan;22(1):19-27. doi: 10.1097/ICU.0b013e3283414284. PMID 21088580
- [Background] Hovding G, Natvik C, Sletteberg O. The refractive error after implantation of a posterior chamber intraocular lens. The accuracy of IOL power calculation in a hospital practice. Acta Ophthalmol (Copenh). 1994 Oct;72(5):612-6. doi: 10.1111/j.1755-3768.1994.tb07188.x. PMID 7887161
- [Background] Norrby S. Sources of error in intraocular lens power calculation. J Cataract Refract Surg. 2008 Mar;34(3):368-76. doi: 10.1016/j.jcrs.2007.10.031. PMID 18299059
- [Background] Norregaard JC, Thoning H, Bernth-Petersen P, Andersen TF, Javitt JC, Anderson GF. Risk of endophthalmitis after cataract extraction: results from the International Cataract Surgery Outcomes study. Br J Ophthalmol. 1997 Feb;81(2):102-6. doi: 10.1136/bjo.81.2.102. PMID 9059242
- [Background] Powell SK, Olson RJ. Incidence of retinal detachment after cataract surgery and neodymium: YAG laser capsulotomy. J Cataract Refract Surg. 1995 Mar;21(2):132-5. doi: 10.1016/s0886-3350(13)80499-3. PMID 7791051
- [Background] Norregaard JC, Thoning H, Andersen TF, Bernth-Petersen P, Javitt JC, Anderson GF. Risk of retinal detachment following cataract extraction: results from the International Cataract Surgery Outcomes Study. Br J Ophthalmol. 1996 Aug;80(8):689-93. doi: 10.1136/bjo.80.8.689. PMID 8949710
- [Background] Qatarneh D, Mathew RG, Palmer S, Bunce C, Tuft S. The economic cost of posterior capsule tear at cataract surgery. Br J Ophthalmol. 2012 Jan;96(1):114-7. doi: 10.1136/bjo.2010.200832. Epub 2011 Mar 1. PMID 21362773
- [Background] Chatoux O, Touboul D, Buestel C, Balcou P, Colin J. [Crystalline lens photodisruption using femtosecond laser: experimental study]. J Fr Ophtalmol. 2010 Sep;33(7):472-80. doi: 10.1016/j.jfo.2010.06.008. French. PMID 20817344
- [Background] Friedman NJ, Palanker DV, Schuele G, Andersen D, Marcellino G, Seibel BS, Batlle J, Feliz R, Talamo JH, Blumenkranz MS, Culbertson WW. Femtosecond laser capsulotomy. J Cataract Refract Surg. 2011 Jul;37(7):1189-98. doi: 10.1016/j.jcrs.2011.04.022. PMID 21700099
- [Background] Palanker DV, Blumenkranz MS, Andersen D, Wiltberger M, Marcellino G, Gooding P, Angeley D, Schuele G, Woodley B, Simoneau M, Friedman NJ, Seibel B, Batlle J, Feliz R, Talamo J, Culbertson W. Femtosecond laser-assisted cataract surgery with integrated optical coherence tomography. Sci Transl Med. 2010 Nov 17;2(58):58ra85. doi: 10.1126/scitranslmed.3001305. PMID 21084720
- [Background] Masket S, Sarayba M, Ignacio T, Fram N. Femtosecond laser-assisted cataract incisions: architectural stability and reproducibility. J Cataract Refract Surg. 2010 Jun;36(6):1048-9. doi: 10.1016/j.jcrs.2010.03.027. No abstract available. PMID 20494782
- [Background] Taketani F, Matuura T, Yukawa E, Hara Y. Influence of intraocular lens tilt and decentration on wavefront aberrations. J Cataract Refract Surg. 2004 Oct;30(10):2158-62. doi: 10.1016/j.jcrs.2004.02.072. PMID 15474830
- [Background] Nagy Z, Takacs A, Filkorn T, Sarayba M. Initial clinical evaluation of an intraocular femtosecond laser in cataract surgery. J Refract Surg. 2009 Dec;25(12):1053-60. doi: 10.3928/1081597X-20091117-04. PMID 20000286
- [Derived] Benard A, Sitta R, Brezin AP, Cochener B, Monnet D, Denis P, Pisella PJ, Hayes N, Schweitzer C; FEMCAT Study Group. Cost Utility and Value of Information Analysis of Femtosecond Laser-Assisted Cataract Surgery. JAMA Ophthalmol. 2023 Jul 1;141(7):625-629. doi: 10.1001/jamaophthalmol.2023.1716. PMID 37200037
- [Derived] Schweitzer C, Brezin A, Cochener B, Monnet D, Germain C, Roseng S, Sitta R, Maillard A, Hayes N, Denis P, Pisella PJ, Benard A; FEMCAT study group. Femtosecond laser-assisted versus phacoemulsification cataract surgery (FEMCAT): a multicentre participant-masked randomised superiority and cost-effectiveness trial. Lancet. 2020 Jan 18;395(10219):212-224. doi: 10.1016/S0140-6736(19)32481-X. PMID 31954466
- [Derived] Schweitzer C, Hayes N, Brezin A, Cochener B, Denis P, Pisella PJ, Benard A; FEMCAT study group. Re: Abell et al.: Cost-effectiveness of femtosecond laser-assisted cataract surgery versus phacoemulsification cataract surgery (Ophthalmology 2014;121:10-6). Ophthalmology. 2014 Oct;121(10):e53-4. doi: 10.1016/j.ophtha.2014.05.025. Epub 2014 Jun 26. No abstract available. PMID 24974812